CLINICAL TRIAL: NCT06732141
Title: Remote Management Strategies and Adherence Improvement for Anxiety-related ICS Resistance in Asthma Patients: an Open-label, Multicenter, Randomized Controlled Trial
Brief Title: Remote Anxiety Management for ICS-resistant Asthma Study
Acronym: RAMICS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Ningbo University (Network)
Responsible Party: Principal Investigator, Chao Cao, Ph.D., Principal Investigator, First Affiliated Hospital of Ningbo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-141A-02
Record Dates: First submitted 2024-12-09; First posted 2024-12-13 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized telephone-based psychological support (Experimental): Participants in this group will receive weekly, personalized 30-minute telephone sessions for 8 weeks, including medication education, lung rehabilitation guidance, motivational interviewing (MI), and progressive muscle relaxation (PMR).
  Interventions: Behavioral: Personalized Telephone-Based Psychological Support
- Standard Care with Weekly Follow-Up Calls (Placebo Comparator): Participants in this group will receive weekly standard care calls for 8 weeks, focusing on health status, asthma symptoms, and medication use, without psychological or educational interventions.
  Interventions: Behavioral: Standard Care with Weekly Follow-Up Calls

INTERVENTIONS:
Behavioral: Personalized Telephone-Based Psychological Support — This intervention involves weekly, individualized 30-minute telephone sessions conducted over 8 weeks. The sessions are designed to address anxiety and improve adherence to inhaled corticosteroid (ICS) therapy in asthma patients. The intervention comprises four core components:
  1. Medication Education: Detailed guidance on the benefits, mechanisms, and safety of ICS therapy, aiming to address misconceptions and reduce fears about side effects.
  2. Lung Rehabilitation Guidance: Instructions for breathing exercises and tailored physical activity to improve respiratory health and overall well-being.
  3. Motivational Interviewing (MI): A patient-centered approach that identifies barriers to adherence, enhances self-efficacy, and motivates behavior change.
  4. Progressive Muscle Relaxation (PMR): A systematic relaxation technique to alleviate physical and emotional stress, tailored to each patient's anxiety levels.
  Arms: Personalized telephone-based psychological support
Behavioral: Standard Care with Weekly Follow-Up Calls — Participants receive weekly telephone follow-up calls for 8 weeks. These calls include health status assessments, symptom monitoring, and general medication inquiries but exclude psychological or educational components.
  Arms: Standard Care with Weekly Follow-Up Calls

SUMMARY:
This study, the Remote Anxiety Management for ICS-resistant Asthma Study (RAMICS), explores strategies to improve medication adherence and anxiety management in asthma patients who are resistant to using inhaled corticosteroids (ICS) due to anxiety. Asthma is a chronic respiratory disease affecting millions worldwide, and ICS therapy is essential for controlling symptoms and preventing severe exacerbations. However, many patients struggle with adherence, especially those with anxiety about ICS side effects. RAMICS is a multicenter, open-label, randomized controlled trial designed to evaluate the effectiveness of personalized telephone-based interventions, including medication education, progressive muscle relaxation (PMR), motivational interviewing (MI), and lung rehabilitation guidance. The study will enroll 216 adult asthma patients with poor ICS adherence and clinically significant anxiety. Participants will be randomized into two groups: the intervention group, receiving weekly telephone sessions, and the control group, receiving standard follow-up calls. The study aims to assess improvements in ICS adherence, reductions in anxiety and depression, better asthma symptom control, and enhanced quality of life. Outcomes will be evaluated immediately after the 8-week intervention and during a 3-month follow-up. By addressing both psychological and medication adherence challenges, this research aims to provide practical solutions for improving asthma management.

ELIGIBILITY:
Inclusion Criteria:

1. Age Requirement:

   Participants must be aged 18 to 80 years, ensuring they are adults capable of making decisions and responding effectively to interventions.
2. Diagnosed Asthma:

   1. Diagnosis must meet the criteria of the Global Initiative for Asthma (GINA) or the American Academy of Asthma guidelines, with at least one confirmed diagnosis by a specialist in the past six months.
   2. Asthma severity must range from mild to moderate persistent, in the chronic management phase, excluding patients in acute exacerbation phases for clearer evaluation of adherence and intervention effects.
3. ICS Treatment History:

   1. Participants must have been on inhaled corticosteroid (ICS) therapy for at least six months, ensuring sufficient treatment history for adherence and effect evaluation.
   2. No major changes to asthma control medication regimen in the past six months, ensuring adherence and intervention outcomes are not confounded by treatment changes.
4. Poor Medication Adherence:

   Identified using the Medication Adherence Report Scale (MARS-10), with an average score <4.5, indicating suboptimal adherence.
5. Presence of Anxiety Symptoms:

   1. Confirmed through the Hamilton Anxiety Rating Scale (HAMA), with a score ≥14, indicating clinically significant anxiety.
   2. Anxiety symptoms must be related to asthma treatment, particularly concerns about ICS side effects or long-term use, ensuring the psychological intervention targets relevant issues.
6. Ability to Communicate by Phone:

   Participants must have stable access to a phone and be willing to engage in telephone-based psychological interventions.
7. Stable Health Condition:

Asthma status must be stable, with no acute exacerbations or significant changes in the past month.

Exclusion Criteria:

1. Severe Psychiatric or Cognitive Disorders:

   1. Diagnosis of major psychiatric disorders, such as major depressive disorder, bipolar disorder, schizophrenia, or other severe mental illnesses within the past six months, based on DSM-5 criteria.
   2. Presence of cognitive impairments or neurological conditions, such as dementia or post-stroke complications, that may affect comprehension or adherence to the intervention.
   3. Current psychiatric treatment involving antipsychotics, antidepressants, or sedatives that could interfere with the intervention's outcomes.
2. Substance Abuse or Dependence:

   History of alcohol or drug abuse within the past six months, including but not limited to opioids, benzodiazepines, or illicit substances.
3. Severe Comorbidities:

   1. Uncontrolled respiratory or cardiovascular conditions, such as chronic obstructive pulmonary disease (COPD), bronchiectasis, interstitial lung disease, heart failure, or uncontrolled hypertension, that could significantly impact asthma control and overall health.
   2. Chronic diseases requiring long-term systemic corticosteroid therapy, such as rheumatic or autoimmune diseases, that may interfere with ICS treatment and study outcomes.
4. Pregnancy or Lactation:

   Pregnant or breastfeeding women are excluded due to the unclear risks of ICS treatment and anxiety management interventions in these populations.
5. Allergic Bronchopulmonary Aspergillosis (ABPA) or Related Conditions:

   Diagnosed ABPA or other respiratory diseases with mechanisms distinct from asthma, which could confound the assessment of ICS treatment effects.
6. Participation in Other Interventional Clinical Trials:

   Participation in another interventional clinical trial within the past three months, particularly those involving respiratory diseases or medication adherence management, to avoid confounding effects on outcomes.
7. Incompatibility with Telephone-Based Interventions:

   Inability to reliably receive or engage in telephone-based psychological interventions due to hearing impairments, communication barriers, or other reasons.
8. Adverse Reactions to Psychological Interventions:

   Documented refusal of or adverse reactions to psychological interventions, such as phone-based relaxation or motivational interviewing, that could affect the feasibility and effectiveness of the study.
9. History of Major Surgery or Hospitalization:

History of major surgery or hospitalization (unrelated to asthma) within the past six months that might impact current health status and introduce bias into the study outcomes.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
ICS Adherence | Baseline, Week 4 (mid-intervention), Week 8 (end of intervention), and 3-month follow-up.
  Medication adherence will be assessed using the Medication Adherence Report Scale (MARS-10), a validated questionnaire. The scale includes 10 items, each scored from 1 (always) to 5 (never), with total scores ranging from 10 to 50. Higher scores indicate better adherence, and a mean score of ≥4.5 reflects good adherence.

SECONDARY OUTCOMES:
Anxiety Levels | Baseline, Week 4 (mid-intervention), Week 8 (end of intervention), and 3-month follow-up.
  Anxiety symptoms will be assessed using the Hamilton Anxiety Rating Scale (HAMA), a validated scale with scores ranging from 0 to 56, where higher scores indicate greater anxiety severity. The intervention aims to reduce anxiety related to ICS use through techniques such as progressive muscle relaxation (PMR) and motivational interviewing (MI).
Depression Levels | Baseline, Week 4 (mid-intervention), Week 8 (end of intervention), and 3-month follow-up.
  Depressive symptoms will be observed using the Hamilton Depression Rating Scale (HAMD), which scores from 0 to 52, with higher scores indicating more severe depression. While the intervention may indirectly impact depressive symptoms, its specific effect on depression is not a primary focus and will require further investigation.
Asthma Control Levels | Baseline, Week 4 (mid-intervention), Week 8 (end of intervention), and 3-month follow-up.
  Asthma symptom control will be assessed using the Asthma Control Test (ACT), a validated questionnaire with scores ranging from 5 to 25. Higher scores indicate better asthma control. The intervention aims to improve asthma control by enhancing ICS adherence and addressing anxiety-related barriers.
Asthma-Related Quality of Life | Baseline, Week 4 (mid-intervention), Week 8 (end of intervention), and 3-month follow-up.
  Health-related quality of life will be evaluated using the Asthma Quality of Life Questionnaire (AQLQ), which measures the impact of asthma on daily activities, social interactions, and overall health perception. The scores range from 1 to 7, with higher scores indicating a better quality of life. The intervention aims to enhance patients' ability to manage asthma and reduce its negative impact on their quality of life.
Incidence of Serious Adverse Events (SAEs) | Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, and 3-month follow-up.
  The safety of the intervention will be assessed by monitoring and recording the incidence of treatment-emergent serious adverse events (SAEs) using the Serious Adverse Event Report Form (SAE Report). The research team will document, analyze, and provide appropriate medical responses to any incidents related to the intervention.
Intervention Adherence | Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8.
  Intervention adherence will be assessed using the Intervention Participation Record, documenting whether participants complete each scheduled telephone session. For the intervention group, adherence to weekly components such as medication education, PMR, and MI will be tracked. For the control group, participation in routine follow-up calls will be recorded.
Asthma Exacerbation Events | Week 4 (mid-intervention), Week 8 (end of intervention), and 3-month follow-up.
  Asthma exacerbation events will be assessed using the Asthma Exacerbation Record, documenting the time, frequency, and severity of each episode. Severity will be graded as mild, moderate, or severe based on international asthma management guidelines. The intervention's effectiveness in reducing exacerbation events will be analyzed.
Frequency of Emergency Department Visits | Week 4 (mid-intervention), Week 8 (end of intervention), and 3-month follow-up.
  The number of emergency department visits due to asthma exacerbations will be tracked using patient self-reports and verified through medical records. This measure assesses the effectiveness of the intervention in reducing the reliance on acute emergency care.
Frequency of Hospitalizations | Week 4 (mid-intervention), Week 8 (end of intervention), and 3-month follow-up.
  The number of hospital admissions due to asthma exacerbations will be documented, including details such as length of stay and treatments administered. This outcome evaluates the intervention's impact on reducing the necessity for inpatient care.
Occurrence of Respiratory Failure | Week 4 (mid-intervention), Week 8 (end of intervention), and 3-month follow-up.
  Documentation of respiratory failure events during hospital stays, including clinical criteria for diagnosis and management details.
Use of Non-Invasive Ventilation | Week 4 (mid-intervention), Week 8 (end of intervention), and 3-month follow-up.
  Documentation of the use of non-invasive ventilation during hospitalization, including indications and duration of use.
ICU Admission and Intubation | Week 4 (mid-intervention), Week 8 (end of intervention), and 3-month follow-up.
  Records of ICU admissions and whether intubation was required during hospitalization, including associated clinical details.
Systemic Steroid Use | Week 4 (mid-intervention), Week 8 (end of intervention), and 3-month follow-up.
  Documentation of systemic corticosteroid use during hospital stays, including dosage and duration.
Length of Hospital Stay | Week 4 (mid-intervention), Week 8 (end of intervention), and 3-month follow-up.
  Total duration of each hospital stay will be recorded to assess the impact of the intervention on hospitalization length.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Second Affiliated Hospital of Harbin Medical University, Harbin
  - Anhui Chest Hospital, Hefei
  - Jingzhou Central Hospital, Jingzhou
  - The First Affiliated Hospital of Ningbo University, Ningbo

IPD SHARING:
Plan to Share IPD: No